CLINICAL TRIAL: NCT01738386
Title: Challenges of Living With Frontotemporal Dementia: The Perspective of the Affected Individual
Brief Title: Living With Frontotemporal Dementia
Status: Terminated | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912153; 12-HG-N153
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2016-02-24

CONDITIONS: Adaptation
Keywords: Adaptation; Coping; Presenile Dementia; Caregiver Burden
MeSH Terms: conditions — Alzheimer Disease; Caregiver Burden

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Background:

- Frontotemporal dementia (FTD) is the second most common cause of early-onset dementia. Alzheimer s disease is the most common. Alzheimer s disease happens most often in the elderly, but FTD typically appears between 40 and 60 years of age. It also has a strong genetic component: Up to 40% of FTD cases are linked to positive family histories. Earlier diagnoses and genetic tests mean that people with FTD will spend more years in earlier stages of disease, aware that they have it. However, few studies have looked at the personal experiences or coping styles of people with FTD. Researchers want to interview people with FTD and their caregivers to understand their experiences with the disease. This information will help create better treatments and therapies for those affected by FTD.

Objectives:

- To study the experiences of persons with FTD and their primary caregivers.

Eligibility:

* Individuals at least 18 years of age who have been diagnosed with FTD.
* Primary caregivers (spouse or partner at least 18 years of age) of individuals who have been diagnosed with FTD.

Design:

* Before FTD participants are recruited, a pilot study will test the interview questions. This pilot study will be given to people with Alzheimer s disease and their caregivers. It will study how well people with dementia understand the interview questions.
* FTD study participants will be recruited through dementia care centers.
* All participants will have in-person interviews. These interviews will take up to 1 hour.
* Participants with FTD will answer questions about their experience with the disease. They will talk about their mental abilities, challenges, and coping strategies.
* Caregivers will answer questions about their experience in caring for someone with FTD. They will talk about their challenges and coping strategies. They will also talk about the person with FTD, and how aware they believe that the person is of the dementia symptoms.
* All participants will receive a small gift card as compensation for their time.
* No treatment will be provided as part of this study.

DETAILED DESCRIPTION:
The purpose of the proposed study is to qualitatively explore the experience, conceptualization of disease, and coping strategies of persons with frontotemporal dementia (FTD). FTD is the second most prevalent cause of early-onset dementia after Alzheimer disease, and has a significant genetic origin. Currently, there are no published studies describing the personal experience or coping styles of individuals with FTD. To accomplish the study s objectives, semi-structured interviews will be conducted with 20 to 30 dyads of patients with FTD and their spouse/partner caregivers. The caregivers will be interviewed about the experience of the person with FTD. Both sets of interviews will be audiotaped, transcribed and subjected to thematic content analysis. Themes emerging in both members of each dyad will be compared and contrasted in order to understand the subjective experience of the disease. Insight into the personal illness experiences of individuals with FTD will inform future clinical intervention studies.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

Participants with FTD must:

* Be affected with any variant of frontotemporal dementia and have documented cognitive impairment
* Have this diagnosis made by a behavioral neurologist, neuropsychologist, psychiatrist, or a group consensus of any of the above in a specialized dementia center

  * For patients recruited through the contact physicians at Johns Hopkins Hospital, University of Pennsylvania, or Columbia University Medical Center, this diagnosis will be verified through personal communication between the interviewer (WM) and the contact physician and through the patients medical records.
  * For patients recruited through a foundation, patient support group or Clinicaltrials.gov, the patients listed dementia care specialist will be contacted to verify the diagnosis, or the appropriate documents obtained through a release of medical information form.
* Be assessed to be in the none (1) to mild (2) impairment category on the Dementia Disability Rating. The assessment must be performed by a dementia care specialist with a medical degree.
* Have an onset of disease at or more than three months before the interview date. This date may or may not differ from the actual date of diagnosis.
* Pass the consent comprehension assessment
* Be 18 or older and speak fluent English

Caregivers participants must:

* Be a spouse or partner who provides day-to-day care for the affected individual.
* Spend a minimum of 16 hours per week, on average in a month, in direct contact with the affected individual.
* NOT be a non-spousal relative, friend, healthcare provider, or hired help.
* Pass the consent comprehension assessment
* Be 18 or older and speak fluent English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-06-13; Study Completion 2016-02-24

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (3):
- United States (3):
  - Johns Hopkins University, Baltimore, Maryland
  - Columbia University, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Ablitt A, Jones G, Muers J. Awareness of carer distress in people with dementia. Int J Geriatr Psychiatry. 2010 Dec;25(12):1246-52. doi: 10.1002/gps.2461. PMID 20033903
- [Background] Baldelli MV, Pirani A, Motta M, Abati E, Mariani E, Manzi V. Effects of reality orientation therapy on elderly patients in the community. Arch Gerontol Geriatr. 1993 Nov-Dec;17(3):211-8. doi: 10.1016/0167-4943(93)90052-j. PMID 15374320
- [Background] Bates J, Boote J, Beverley C. Psychosocial interventions for people with a milder dementing illness: a systematic review. J Adv Nurs. 2004 Mar;45(6):644-58. doi: 10.1046/j.1365-2648.2003.02959.x. PMID 15012642